CLINICAL TRIAL: NCT02616861
Title: A 2-stage Phase 1 Study of Safety, Tolerability, PK, and PD of IW-1973 Tablet in Healthy Volunteers in an Open-label, Single-dose Stage, and a Randomized, Double Blind, Placebo-controlled, Multiple-ascending-dose Stage
Brief Title: Trial of IW-1973 (A Stimulator of Soluble Guanylate Cyclase (sGC)) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cyclerion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICP-1973-102
Record Dates: First submitted 2015-10-29; First posted 2015-11-30 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — praliciguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IW-1973 (Experimental): 1973 Escalating Doses
  Interventions: Drug: IW-1973
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Matching Placebo Tablet

INTERVENTIONS:
Drug: IW-1973 — IW-1973 Tablet
  Arms: IW-1973
Drug: Matching Placebo Tablet — Matching placebo tablet
  Arms: Placebo

SUMMARY:
Stage 1: To assess the safety, tolerability, pharmacokinetic (PK) profile, and pharmacodynamic (PD) effects of the IW-1973 Tablet administered orally to healthy volunteers, in fed and fasted states, in a single-dose crossover study.

Stage 2: To assess the safety, tolerability, PK profile, and PD effects of a range of doses of IW-1973 Tablet administered orally to healthy subjects in a 21-day, multiple ascending-dose study with optional up-titration of dose level within cohort.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an ambulatory male or female between 18 and 55 years old at the Screening Visit
* Subject's body mass index score is > 18.5 and < 30.0 kg/m2 at the Screening Visit
* Women of childbearing potential must have a negative pregnancy test and must agree to use double-barrier contraception
* Subject is in good health and has no clinically significant findings on a physical examination
* Other inclusion criteria per protocol

Exclusion Criteria:

* History of any clinically significant medical condition
* Other exclusion criteria per protocol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events | 42 Days
Maximum observed plasma concentration (Cmax) | 42 Days
Blood Pressure | 42 days
Area under the plasma concentration time curve during a dosing interval (AUC) | 42 Days
Time of maximum observed plasma concentration (Tmax) | 42 Days
Heart rate | 42 Days
Serum cGMP | 42 Days

CONTACTS AND LOCATIONS:
Overall Officials: John Hanrahan, MD, Study Director — Ironwood Pharmaceuticals
Locations (1):
- Ironwood Investigator, San Antonio, Texas, United States